CLINICAL TRIAL: NCT03594591
Title: Changes in the Retinal and Carotid Microcirculation After Restoring Normoglycemia in Patients With Type 2 Diabetes (OCTAUS-T2D Study)
Brief Title: Changes in the Retinal and Carotid Microcirculation After Restoring Normoglycemia in Patients With Type 2 Diabetes
Acronym: OCTAUS-T2D
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other)
Responsible Party: Principal Investigator, Emilio Ortega Martínez de Victoria, Principal Investigator, Consultant Endocrinologist, Hospital Clinic of Barcelona
Other Study IDs: PI 17/01479
Record Dates: First submitted 2018-05-10; First posted 2018-07-20 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes Mellitus; Microangiopathy; Diabetic Retinopathy; Arteriosclerosis; Carotid Atherosclerosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Retinopathy; Arteriosclerosis; Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Antidiabetic treatment by usual care — Observation of changes in the microcirculation after optimization of antidiabetic therapy by usual care.

SUMMARY:
This is a prospective and observational study in patients with type two diabetes. The study hypothesis is that chronic hyperglycemia causes an increase in the microcirculation on the carotid artery wall and retina, evaluated by angio-OCT. Furthermore, the reestablishment of normoglycemia would decrease this microcirculation, which could trigger hypoxic and ischemic changes, accelerating preclinical atherosclerosis. The study goal is to describe the microangiopathy in both territories in patients with type two diabetes and chronic hyperglycemia, and to evaluate changes after the reestablishment of normoglycemia.

DETAILED DESCRIPTION:
This is a prospective and observational study in patients with type two diabetes. The study hypothesis is that chronic hyperglycemia causes an increase in the microcirculation on the carotid artery wall (evaluating vasa vasorum by contrast-assessed carotid ultrasound) and retina (evaluated by angio-OCT). Furthermore, the reestablishment of normoglycemia would decrease this microcirculation, which could trigger hypoxic and ischemic changes, accelerating preclinical atherosclerosis. The primary outcome is to describe the microangiopathy in both territories in 20 patients with type two diabetes and chronic hyperglycemia (basal), and to evaluate the changes after the reestablishment of normoglycemia (at 1, 3 and 6 months). Additionally, clinical, laboratory, diet and biomarkers will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type two diabetes with chronic hyperglycemia (HbA1c >9%) in who a swift and maintained improvement in glycemic control is expected, as a consequence of the antidiabetic treatment decided by usual care owing to the clinical situation.

   This treatment will include, in many cases, albeit not always, insulin (basal, basal-plus, mixes, or multiple doses). The usual clinical scenario will be failure to non-insulin antidiabetic drugs or to combined treatment (basal insulin and non-insulin drugs). Patients with new diagnose of type two diabetes who start treatment (insulin and non-insulin drugs) in which a long-evolution diabetes is suspected will also be candidates.
2. Caucasian and age between 35 and 75 years.
3. Informed consent by the patient or legal tutor.

Exclusion Criteria:

1. Previous history of carotid territory interventionism (stent o endarterectomy).
2. Presence of carotid plaques in the first centimetre of the posterior wall of the common carotid artery.
3. Ophtalmologic: Proliferative diabetic retinopathy and/or diabetic macular oedema, retinal photocoagulation, intravitreous therapy and/or vitreo-retinal surgery, myopia of >6 diopters, history of non-diabetic vascular retinopathy.
4. Stage 4 chronic kidney disease (estimated glomerular filtration <30 ml/min/1,73m2), organ transplant, HIV chronic infection, active tuberculosis, active malaria, chronic b or C hepatitis, cirrhosis or intestinal inflammatory disease.
5. Current pregnancy or breastfeeding, o gestational desire in the following two years.
6. History of alcohol or drug dependence (except for caffeine and nicotine) in the former 5 years, active depression or psychiatric disease, dementia, presence of another chronic or debilitating disease with short life-expectancy, institutionalization or severe disability.
7. Presence of contraindications for the use of ecographic contrast.
8. Current Participation in another study protocol.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type two diabetes with chronic hyperglycemia (HbA1c >9%) in who a swift and maintained improvement in glycemic control is expected, as a consequence of the antidiabetic treatment decided by usual care owing to the clinical situation. Patients with new diagnose of type two diabetes who start treatment (insulin and non-insulin drugs) in which a long-evolution diabetes is suspected will also be candidates.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes in retinal microcirculation (perifoveal vessel density) | 0, 1, 3 and 6 months
  Changes in perifoveal vessel density, OCTA images will be processed to obtain vascular density measurements in this area (mm-1)
Changes in arterial wall microcirculation (vasa-vasorum density) | 0, 3 and 6 months
  Changes vasa-vasorum (VV) density, VV signal as the ratio of the contrast agent signal of the VV and that of the lumen of the artery

SECONDARY OUTCOMES:
Changes in retinal microcirculation (Parafoveal vessel density ) | 0, 1, 3 and 6 months
  OCTA images will be processed to obtain vascular density measurements in this area (mm-1)
Changes in retinal microcirculation (Total Avascular Area ) | 0, 1, 3 and 6 months
  OCTA images will be processed to obtain total avascular area measurements (mm2)
Changes in retinal microcirculation (Foveal Avascular Area) | 0, 1, 3 and 6 months
  OCTA images will be processed to obtain foveal avascular zone area measurements (mm2)

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Ortega, MD; PhD, Principal Investigator — Hospital Clínic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Action to Control Cardiovascular Risk in Diabetes Study Group; Gerstein HC, Miller ME, Byington RP, Goff DC Jr, Bigger JT, Buse JB, Cushman WC, Genuth S, Ismail-Beigi F, Grimm RH Jr, Probstfield JL, Simons-Morton DG, Friedewald WT. Effects of intensive glucose lowering in type 2 diabetes. N Engl J Med. 2008 Jun 12;358(24):2545-59. doi: 10.1056/NEJMoa0802743. Epub 2008 Jun 6. PMID 18539917
- [Background] Sanahuja J, Alonso N, Diez J, Ortega E, Rubinat E, Traveset A, Alcubierre N, Betriu A, Castelblanco E, Hernandez M, Purroy F, Arcidiacono MV, Jurjo C, Fernandez E, Puig-Domingo M, Groop PH, Mauricio D. Increased Burden of Cerebral Small Vessel Disease in Patients With Type 2 Diabetes and Retinopathy. Diabetes Care. 2016 Sep;39(9):1614-20. doi: 10.2337/dc15-2671. Epub 2016 Jun 8. PMID 27281772
- [Background] Arcidiacono MV, Rubinat E, Borras M, Betriu A, Trujillano J, Vidal T, Mauricio D, Fernandez E. Left carotid adventitial vasa vasorum signal correlates directly with age and with left carotid intima-media thickness in individuals without atheromatous risk factors. Cardiovasc Ultrasound. 2015 Apr 17;13:20. doi: 10.1186/s12947-015-0014-7. PMID 25889409
- [Background] Catalan M, Herreras Z, Pinyol M, Sala-Vila A, Amor AJ, de Groot E, Gilabert R, Ros E, Ortega E. Prevalence by sex of preclinical carotid atherosclerosis in newly diagnosed type 2 diabetes. Nutr Metab Cardiovasc Dis. 2015 Aug;25(8):742-8. doi: 10.1016/j.numecd.2015.04.009. Epub 2015 May 7. PMID 26033395
- [Background] Dimitrova G, Chihara E, Takahashi H, Amano H, Okazaki K. Author Response: Quantitative Retinal Optical Coherence Tomography Angiography in Patients With Diabetes Without Diabetic Retinopathy. Invest Ophthalmol Vis Sci. 2017 Mar 1;58(3):1767. doi: 10.1167/iovs.17-21706. No abstract available. PMID 28334376